CLINICAL TRIAL: NCT04113590
Title: Laparoscopic Assisted Transvaginal Cholecystecomy
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: no patients were enrolled
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: STU 122010-059
Record Dates: First submitted 2012-07-03; First posted 2019-10-03 (Actual); Last update posted 2019-10-03 (Actual); Status verified 2019-10

CONDITIONS: Cholelithiasis
Keywords: cholecystectomy; gall stone surgery; scarless surgery; cholelithiasis
MeSH Terms: conditions — Cholelithiasis | interventions — Cholecystectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Transvaginal cholecystectomy under laparoscopic guidance (Experimental): The removal of the gallbladder through several small incisions using a camera to see is called laparoscopic cholecystectomy. This study is being done to evaluate whether cholecystectomy can be performed through a natural orifice (the vagina) with minimal laparoscopic assistance (only one abdominal trocar versus four in the routine laparoscopic cholecystectomy).
  Interventions: Procedure: Laparoscopic Assisted Transvaginal Cholecystectomy

INTERVENTIONS:
Procedure: Laparoscopic Assisted Transvaginal Cholecystectomy — Perform transvaginal cholecystectomy while obtaining safe access under laparoscopic visualization
  Other Names: Transvaginal (TV) NOTES; scarless cholecystectomy; cholecystectomy

SUMMARY:
Laparoscopic cholecystectomy is currently the standard procedure for removing the gallbladder. This procedure usually requires the insertion of four trocars into the abdomen for passage of laparoscopic instruments; each trocar requires a small incision, which results in postoperative pain and scarring. There has recently been a tremendous surge in interest within the surgical community to further reduce the pain, invasiveness, and cosmesis of laparoscopic surgery. To achieve this goal, surgeons are either reducing the number of trocars placed through the abdominal wall or eliminating them completely The goal of this project is to evaluate the feasibility of performing transvaginal cholecystectomy while obtaining safe access under laparoscopic visualization. This has the potential to decrease postoperative pain, improve cosmesis, and lead to a shorter recovery following cholecystectomy.

DETAILED DESCRIPTION:
20 female patients will be enrolled. Patients who are scheduled to undergo elective laparoscopic cholecystectomy will be invited to participate in this study. The laparoscopic instrumentation will be sterilized using standard methods. Conventional and new laparoscopic and endoscopic equipment will be used for this project; all equipment is commercially available and is FDA-approved for laparoscopic procedures. Access will be obtained into the peritoneal cavity at the umbilicus in a standard fashion, either by use of a Veress needle technique or by insertion of a trocar using the open technique. Through a single umbilical incision, a 5mm trocar will be placed into the peritoneal cavity. A 5mm laparoscope will then be inserted into the peritoneal cavity. This will be used to monitor safe peritoneal entry of a dilating12mm transvaginal trocar. Subsequent operative visualization will be by use of a flexible endoscope which will be placed through the transvaginal port. The gallbladder will be retracted using sutures as well as endoscopic and / or laparoscopic graspers. In order to obtain the critical view of safety [5] the cystic duct and artery will be dissected, ligated and divided by use of conventional laparoscopic and new articulating instruments. The dissected gallbladder will be retrieved transvaginally. If for any reason suitable retraction or dissection cannot be performed using the transvaginal strategy, the case will be promptly converted to a standard laparoscopic approach by the insertion of additional transabdominal trocars.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled to undergo elective laparoscopic cholecystectomy
* Women 18-75 years of age
* English or Spanish speaking

Exclusion Criteria:

* American Society of Anesthesiologists (ASA) classification of ≥ 3
* Morbid obesity (BMI ≥35)
* Pregnant women
* Acute cholecystitis
* Any ongoing intra-abdominal infection
* Prior upper abdominal or pelvic surgery and/or adhesions
* Virgins
* Women with an active sexually transmitted disease or any vaginal infection
* History of dyspareunia

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-08; Primary Completion 2012-12 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] using a Quality of Life scale | 23 hours post op
  The primary outcome of this study will be to evaluate the feasibility of performing a transvaginal cholecystectomy while obtaining safe access under laparoscopic visualization. A postoperative Quality of Life questionnaire will be given to the patient to access pain. We will also address whether cosmesis was a factor for their decision. Operative time will be tracked as well as standard operative outcomes including any complications. Patients will be kept for 23 hours observation postoperatively and will follow up in the clinic.
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] using a Visual Analog Scale | 23 hours post op
  The primary outcome of this study will be to evaluate the feasibility of performing a transvaginal cholecystectomy while obtaining safe access under laparoscopic visualization. A Visual Analog Scale for pain will be given to the patient to access pain. We will also address whether cosmesis was a factor for their decision. Operative time will be tracked as well as standard operative outcomes including any complications. Patients will be kept for 23 hours observation postoperatively and will follow up in the clinic.The Visual Analog Scale is a scale from 0-10, with 10 being a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Scott, MD, Principal Investigator — UT Southwestern

REFERENCES:
- [Background] Scott DJ, Tang SJ, Fernandez R, Bergs R, Goova MT, Zeltser I, Kehdy FJ, Cadeddu JA. Completely transvaginal NOTES cholecystectomy using magnetically anchored instruments. Surg Endosc. 2007 Dec;21(12):2308-16. doi: 10.1007/s00464-007-9498-z. Epub 2007 Aug 18. PMID 17704871
- [Background] Zorron R, Maggioni LC, Pombo L, Oliveira AL, Carvalho GL, Filgueiras M. NOTES transvaginal cholecystectomy: preliminary clinical application. Surg Endosc. 2008 Feb;22(2):542-7. doi: 10.1007/s00464-007-9646-5. Epub 2007 Nov 20. PMID 18027043
- [Background] Elazary R, Khalaileh A, Shussman N, Schlager A, Horgan S, Talamini MA, Rivkind AI, Mintz Y. [Surgery without incisions--the third generation of surgery]. Harefuah. 2011 Jan;150(1):25-8, 69. Hebrew. PMID 21449152
- [Background] Schlager A, Khalaileh A, Shussman N, Elazary R, Keidar A, Pikarsky AJ, Ben-Shushan A, Shibolet O, Horgan S, Talamini M, Zamir G, Rivkind AI, Mintz Y. Providing more through less: current methods of retraction in SIMIS and NOTES cholecystectomy. Surg Endosc. 2010 Jul;24(7):1542-6. doi: 10.1007/s00464-009-0807-6. Epub 2009 Dec 25. PMID 20035352
- [Background] Christian J, Barrier BF, Schust D, Miedema BW, Thaler K. Culdoscopy: a foundation for natural orifice surgery--past, present, and future. J Am Coll Surg. 2008 Sep;207(3):417-22. doi: 10.1016/j.jamcollsurg.2008.01.032. Epub 2008 May 5. No abstract available. PMID 18722948
- [Background] Auyang ED, Santos BF, Enter DH, Hungness ES, Soper NJ. Natural orifice translumenal endoscopic surgery (NOTES((R))): a technical review. Surg Endosc. 2011 Oct;25(10):3135-48. doi: 10.1007/s00464-011-1718-x. Epub 2011 May 7. PMID 21553172